CLINICAL TRIAL: NCT02879851
Title: Evaluation of the Accuracy of the Elastic Fusion MRI-ultrasound ((Magnetic Resonance Imaging) Obtained in Vivo by the Koelis™ System
Brief Title: Evaluation of the Accuracy of the Elastic Fusion MRI-ultrasound Obtained in Vivo by the Koelis™ System
Acronym: EFEL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0422
Record Dates: First submitted 2016-08-09; First posted 2016-08-26 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Cancer of the Prostate
Keywords: ultrasound; Koelis system; MRI; gold grain
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The study aims at quantifying the registration error obtained in routine patients in different parts of the prostate and for operators with different experience in order to assess the average precision of the elastic MR-ultrasound fusion obtained by Koelis™ system.

Patients referred for placement of intraprostatic fiducials before radiotherapy for prostate cancer will be prospectively offered to enter the study.

The fiducials will be placed under transrectal ultrasound guidance, in the prostate apex, midgland and base, according to our routine procedure. A 3D Ultrasound acquisition of the prostate will be obtained at the end of the placement. As per our routine procedure, patients will undergo unenhanced prostate MRI to control the position of the fiducials. An elastic fusion of the MR images and the 3D ultrasound acquisitions will be retrospectively performed by operators of varying experience using the Koelis system. The fiducials (visible on MR and ultrasound images) will be used to quantify the registration error.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient requiring placement of intraprostatic fiducials
* No contra-indication for fiducials placement
* No contra -indication to MRI
* No contra -indication for intravenous injection of gadolinium chelates
* Patient affiliated to the social security system
* Patients who received oral and written information

Exclusion Criteria:

* Patient deprived of liberty as a result of a judicial or administrative decision.
* Patient under guardianship or curatorship.
* Any event preventing or prematurely interrupting the collection of assessment criteria would result in the premature exit of the subject.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with prostate cancer referred for placement of intraprostatic fiducials before prostate radiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the overall registration obtained by the Koelis™ system | 1 month
  The fusion will be performed retrospectively without interfering with patient management. This fusion is an off-line analysis that will be performed within one month of the images acquisition. Each of the four operators will perform a US/MR fusion for all patients and will be blinded to the fusions performed by the others. The results will be presented when all operators have finished the fusions in all patients.
  The overall registration error (TRE3D, defined as the Euclidean distance between the US marker and the MR marker after fusion) will be calculated based on the 3D coordinates of the fiducials on MR and ultrasound images.

SECONDARY OUTCOMES:
Influence on TRE3D of the position of the fiducials (apex, midgland and base) | 1 month
  The fusion will be performed retrospectively without interfering with patient management. This fusion is an off-line analysis that will be performed within one month of the images acquisition. Each of the four operators will perform a US/MR fusion for all patients and will be blinded to the fusions performed by the others. The results will be presented when all operators have finished the fusions in all patients.
  The distribution of TRE3D for the markers at the apex, midgalnd and base will be compared
Influence on TRE3D of the experience of the fusion operators | 1 month
  The fusion will be performed retrospectively without interfering with patient management. This fusion is an off-line analysis that will be performed within one month of the images acquisition. Each of the four operators will perform a US/MR fusion for all patients and will be blinded to the fusions performed by the others. The results will be presented when all operators have finished the fusions in all patients.
  The distribution of TRE3D for the four operators will be compared

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of Edouard Herriot, Lyon, France